CLINICAL TRIAL: NCT04124003
Title: An Open-label, Single-sequence, Drug-drug Interaction Study to Assess the Effect of BMS-963272 Coadministration on the Systemic Exposure of Rosuvastatin in Healthy Participants
Brief Title: A Study to Assess the Drug-drug Interaction of BMS-963272 and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MB006-018
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rosuvastatin + BMS-963272 (Experimental)
  Interventions: Drug: rosuvastatin; Drug: BMS-963272

INTERVENTIONS:
Drug: rosuvastatin — Specified dose on specified days
Drug: BMS-963272 — Specified dose on specified days

SUMMARY:
Phase 1 study that assesses the effect of BMS-963272 on exposure of rosuvastatin in healthy participants

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participants, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Women must not be of childbearing potential (WNOCBP)
* Women and men must agree to follow instructions for methods of contraception

Exclusion Criteria:

* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study.
* Any major surgery within 4 weeks of study drug administration
* Any blood transfusion or donation of blood to a blood bank or in a clinical study within 4 weeks of study drug administration
* Previous treatment with BMS-963272
* Participants who smoke, as well as, those who have stopped smoking less than 6 months prior to day 1

Other protocol-defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | up to Day 10
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration AUC(0-T) | up to Day 10
Area under the plasma concentration-time curve extrapolated to infinity AUC (INF) | up to Day 10

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Approximately 50 days
Number of significant changes in lab assessments of blood serum | Approximately 50 days
Number of significant changes in lab assessments of blood | Approximately 50 days
Number of significant changes in lab assessments of urine | Approximately 50 days
Blood pressure | Approximately 50 days
Body temperature | Approximately 50 days
Respiratory rate | Approximately 50 days
Number of Participants with abnormal physical examination findings | Approximately 50 days
Heart rate | Approximately 50 days
Number of participants with 12-lead Electrocardiogram (ECG) Abnormalities | Approximately 50 days

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences - Salt Lake, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm